CLINICAL TRIAL: NCT03541733
Title: The Bowel Preparation for Magnetic Resonance Enterography: a Open Label, Multicenter Randomized Controlled Trial
Brief Title: Bowel Preparation for Magnetic Resonance Enterography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Collaborators: Wuxi No. 2 People's Hospital (Other)
Responsible Party: Principal Investigator, Faming Zhang, Associate chief physician, associate professor, The Second Hospital of Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MRE-CN-180421
Record Dates: First submitted 2018-05-05; First posted 2018-05-30 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Crohn Disease
Keywords: magnetic resonance enterography; bowel preparation
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tubing-group (Experimental): mid-gut tubing prior to the MRE examination, administer contrast solution through the mid-gut tube
  Interventions: Other: mid-gut tubing
- Oral-group (No Intervention): administer contrast solution orally, mid-gut tubing after the MRE examination

INTERVENTIONS:
Other: mid-gut tubing — mid-gut tubing at different time
  Arms: Tubing-group

SUMMARY:
Adequate bowel preparation is required for magnetic resonance enterography (MRE) which can be achieved by two methods including administering contrast solution after mid-gut tubing and taking contrast solution orally. We present the design of randomized controlled trial to compare the efficacy and compliance of bowel preparation through mid-gut tubing with taking contrast orally for MRE in patients with Crohn's disease (CD).

DETAILED DESCRIPTION:
This is a open label, multicenter, randomized controlled trial. 96 patients are planed to be 1:1 randomized into one of two groups: (1) Tube group, mid-gut tubing prior to the MRE examination, administer contrast solution through the mid-gut tube; (2) Oral group, administer contrast solution orally, mid-gut tubing after the MRE examination. The primary outcome measures are: (1) grade of bowel distention evaluated by a 5-grade scale (1 = 0-20% segmental distention, 2 = 20-40% distention, 3 = 40-60% distention, 4 = 60-80% distention, 5 = 80-100% distention); (2) degree of discomfort before/during/after bowel preparation for MRE using a visual 5-grade to describe the severity of nervousness, nausea, vomiting, bloating, abdominal pain, and diarrhea (1 = few, 5 = very severe). The secondary outcome measure is the accuracy of lesion detection through MRE confirmed by endoscopy (within 1 month before MRE and during this hospitalization) will be evaluated by a 5-point scale (lesions locating at the terminal ileum, ileocecal junction, hepatic flexure of colon, splenic flexure of colon, and rectosigmoid colon, consistency of lesion detection from each bowel segment scoring 1 point, otherwise not scoring).

ELIGIBILITY:
Inclusion Criteria:

* Patients with CD need MRE examination and mid-gut tubing (prepared for fecal microbiota transplantation and/or enteral nutrition);
* Age ≥ 14 years old.

Exclusion Criteria:

* Unable to understand or provide informed consent;
* Had difficulty in swallowing, or dysphagia;
* Allergic to laxative and/or contrast;
* Claustrophobia or implanted metal objects or cardiac pacemaker precluding performance of MRI;
* Known or suspected intestinal obstruction or severe stricture.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
grade of bowel distention | one year
  grade of bowel distention evaluated by a 5-grade scale (1 = 0-20% segmental distention, 2 = 20-40% distention, 3 = 40-60% distention, 4 = 60-80% distention, 5 = 80-100% distention)
degree of discomfort | one year
  using a visual 5-grade to describe the severity of nervousness, nausea, vomiting, bloating, abdominal pain, and diarrhea (1 = few, 5 = very severe)

SECONDARY OUTCOMES:
accuracy of lesion detection | one year
  accuracy of lesion detection through MRE confirmed by endoscopy (within 1 month before MRE and during this hospitalization) will be evaluated by a 5-point scale (lesions locating at the terminal ileum, ileocecal junction, hepatic flexure of colon, splenic flexure of colon, and rectosigmoid colon, consistency of lesion detection from each bowel segment scoring 1 point, otherwise not scoring)

CONTACTS AND LOCATIONS:
Overall Officials: Faming Zhang, MD, PhD, Principal Investigator — The Second Hospital of Nanjing Medical University
Locations (1):
- Fmt-Dt-N-27/1350, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ajaj W, Goehde SC, Schneemann H, Ruehm SG, Debatin JF, Lauenstein TC. Oral contrast agents for small bowel MRI: comparison of different additives to optimize bowel distension. Eur Radiol. 2004 Mar;14(3):458-64. doi: 10.1007/s00330-003-2177-0. Epub 2003 Nov 22. PMID 14634782
- [Background] Cui B, Feng Q, Wang H, Wang M, Peng Z, Li P, Huang G, Liu Z, Wu P, Fan Z, Ji G, Wang X, Wu K, Fan D, Zhang F. Fecal microbiota transplantation through mid-gut for refractory Crohn's disease: safety, feasibility, and efficacy trial results. J Gastroenterol Hepatol. 2015 Jan;30(1):51-8. doi: 10.1111/jgh.12727. PMID 25168749
- [Background] Masselli G, Casciani E, Polettini E, Gualdi G. Comparison of MR enteroclysis with MR enterography and conventional enteroclysis in patients with Crohn's disease. Eur Radiol. 2008 Mar;18(3):438-47. doi: 10.1007/s00330-007-0763-2. Epub 2007 Sep 25. PMID 17899102
- [Background] Negaard A, Paulsen V, Sandvik L, Berstad AE, Borthne A, Try K, Lygren I, Storaas T, Klow NE. A prospective randomized comparison between two MRI studies of the small bowel in Crohn's disease, the oral contrast method and MR enteroclysis. Eur Radiol. 2007 Sep;17(9):2294-301. doi: 10.1007/s00330-007-0648-4. Epub 2007 May 5. PMID 17483955
- [Background] Long C, Yu Y, Cui B, Jagessar SAR, Zhang J, Ji G, Huang G, Zhang F. A novel quick transendoscopic enteral tubing in mid-gut: technique and training with video. BMC Gastroenterol. 2018 Mar 13;18(1):37. doi: 10.1186/s12876-018-0766-2. PMID 29534703
- [Derived] Wang Y, Dai M, Zheng M, Jin Y, Wen Q, Cui B, Zhang Z, Zhu J, Zhang F. Bowel preparation after mid-gut tubing enhanced the efficacy and compliance of magnetic resonance enterography in Crohn's disease: a randomized controlled trial. Therap Adv Gastroenterol. 2024 Sep 26;17:17562848241275337. doi: 10.1177/17562848241275337. eCollection 2024. PMID 39346010
- [Derived] Dai M, Zhang T, Li Q, Cui B, Xiang L, Ding X, Rong R, Bai J, Zhu J, Zhang F. The bowel preparation for magnetic resonance enterography in patients with Crohn's disease: study protocol for a randomized controlled trial. Trials. 2019 Jan 3;20(1):1. doi: 10.1186/s13063-018-3101-x. PMID 30606236